CLINICAL TRIAL: NCT05372276
Title: A Comparison of Mental Toughness and Mental Imagination Skills of Professional Esports Players With Different Levels of Physical Activity
Brief Title: Comparison of Mental Skills of Professional Esports Players With Different Levels of Physical Activity
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gulfidan Tokgoz, Lecturer, Istanbul University - Cerrahpasa
Other Study IDs: Istanbul Universty-Cerrahpasa
Record Dates: First submitted 2022-05-09; First posted 2022-05-12 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2023-05

CONDITIONS: Healthy; Physical Inactivity
Keywords: esport; physical activity; mental toughness; mental imaginery
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Inactive: The score obtained by multiplying the duration, frequency and MET values of the physical activities in which the participants participated in 7 days and for at least 10 minutes is <600 MET - min/week.
  After the participants are divided into groups according to their physical activity levels, mental toughness and mental imagery skills will be evaluated with the Mental Toughness Scale and the Sports Imagery Questionnaire.
  Interventions: Other: Assessment 1; Other: Assessment 2; Other: Assessment 3; Other: Assessment 4
- Low Level Physical Activity (PA): The score obtained by multiplying the duration, frequency and MET values of the physical activities in which the participants participated in 7 days and for at least 10 minutes is 600 - 3000 MET - min/week.
  After the participants are divided into groups according to their physical activity levels, mental toughness and mental imagery skills will be evaluated with the Mental Toughness Scale and the Sports Imagery Questionnaire.
  Interventions: Other: Assessment 1; Other: Assessment 2; Other: Assessment 3; Other: Assessment 4
- Adequate Level Physical Activity (PA): The score obtained by multiplying the duration, frequency and MET values of the physical activities in which the participants participated in 7 days and for at least 10 minutes is >3000 MET - min/week.
  After the participants are divided into groups according to their physical activity levels, mental toughness and mental imagery skills will be evaluated with the Mental Toughness Scale and the Sports Imagery Questionnaire.
  Interventions: Other: Assessment 1; Other: Assessment 2; Other: Assessment 3; Other: Assessment 4

INTERVENTIONS:
Other: Assessment 1 — Mental Toughness Questionnaire in Sport
Other: Assessment 2 — Sport Imagery Questionnaire
Other: Assessment 3 — The Pittsburgh Sleep Quality Index
Other: Assessment 4 — The Perceived Stress Scale (PSS)

SUMMARY:
Competitive video games, defined as esports, have been increasing in popularity especially in the last ten years.

In this study, our primary aim is; to compare the mental abilities of professional esport players with different physical activity levels.

DETAILED DESCRIPTION:
Competitive video games, defined as esports, have been increasing in popularity especially in the last ten years.

In this study, our primary aim is; to compare the mental abilities of professional esport players with different physical activity levels.

The second aim of our study is; to reveal information about the physical activity levels of Turkish professional esports players. In addition, pioneering information will be presented to both clinicians and researchers on physical activity in esports, which is frequently discussed today.

ELIGIBILITY:
Inclusion Criteria:

* Beingover 18 years old
* Being a professional esports player
* Being contracted with an esports club
* Esports branch includes games played on a computer platform, in sitting position, using mouse, keyboard and monitor.
* Volunteering for the study

Exclusion Criteria:

* Sports branches in which different equipments that can change biomechanical properties such as phone, console, joystick are used.
* Having less than 2 years of esports background
* Having any musculoskeletal injury within 6 months
* Having any neurological, rheumatological, cardiac problems
* Having a psychiatric illness
* Having any communication problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample of this research will be formed by professional esports players living in Turkey.
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
The International Physical Activity Questionnaires (IPAQ) | 3 months, July 2022 - September 2022
  The short form of the International Physical Activity Questionnaire (UFAA) will be used to determine the physical activity levels of the participants. The UFAA-Short Form is a valid tool used to assess physical activity in young adults. It is a 7-item scale that evaluates the duration and frequency of vigorous physical activity, moderate physical activity, walking and sedentary behavior based on MET values. Physical activity levels are classified into 3 categories according to the scores obtained by multiplying the duration, frequency and MET values of the physical activities that the participants participated in within 7 days and for at least 10 minutes. Accordingly, <600 MET - min/week is defined as inactive, 600 - 3000 MET - min/week low, and >3000 MET - min/week is defined as sufficient physical activity level.

SECONDARY OUTCOMES:
Mental Toughness Questionnaire in Sports | 4 months, September 2022 - December 2022
  The mental toughness parameters of the participants will be evaluated face-to-face with the Mental Toughness Questionnaire in Sports. It was developed by Sheard, Golby and Van Wersch in 2009. It is a 14-item scale that includes three sub-dimensions of trust, continuity and control and provides information about mental resilience in young adults. Although there are reverse questions in the scale, it includes a Likert-type evaluation between 1 and 4 (1= Completely false, 4= Completely true). Although the highest score that can be obtained is 56, high scores from the scale show that the athletes have a high level of mental endurance.
Sport Imagery Questionaire | 4 months, September 2022 - December 2022
  The imagination skills of the participants will be evaluated face-to-face with the Sports Imagery Questionnaire. It is a 30-item scale developed by Hall, Mack, Paivio, and Hausenblas in 1998, including 5 sub-dimensions. Each item included in the scale is scored between 1 and 7 by the athletes. Although the highest score that can be obtained is 210, high scores indicate an increase in visualization skills.

OTHER OUTCOMES:
The Pittsburgh Sleep Quality Index (PSQI) | 4 months, September 2022 - December 2022
  PUKI is a self-report scale that assesses sleep quality and sleep disturbance over a one-month period. PUKI was published in 1989 by Buysse et al. and it has been shown to have sufficient internal consistency, test-retest reliability and validity. In the evaluation of PUKI, 18 items are included in the scoring. The total score has a value between 0-21, a high total score indicates poor sleep quality. A total PUKI score of ≤5 indicates "good sleep quality", and >5 indicates "poor sleep quality".
The Perceived Stress Scale (PSS) | 4 months, September 2022 - December 2022
  Cohen et al. (1983) was designed to determine how stressful the individual perceives certain situations in his life. There are two short forms of PSS with 10 and 4 items. Scoring of PASS-10 ranges from 0 to 40. A high score indicates an excess of one's perception of stress.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Zengin Alpozgen, PhD, Study Director — Istanbul University - Cerrahpasa; Gulfidan Tokgoz, MSc, Principal Investigator — Istanbul University - Cerrahpasa; Sahra Şirvan Can, MSc, Principal Investigator — Istanbul University - Cerrahpasa; Doğukan Tongar, MsC, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Papathanasiou G, Georgoudis G, Georgakopoulos D, Katsouras C, Kalfakakou V, Evangelou A. Criterion-related validity of the short International Physical Activity Questionnaire against exercise capacity in young adults. Eur J Cardiovasc Prev Rehabil. 2010 Aug;17(4):380-6. doi: 10.1097/HJR.0b013e328333ede6. PMID 19940775
- [Background] Gucciardi DF, Hanton S, Fleming S. Are mental toughness and mental health contradictory concepts in elite sport? A narrative review of theory and evidence. J Sci Med Sport. 2017 Mar;20(3):307-311. doi: 10.1016/j.jsams.2016.08.006. Epub 2016 Aug 9. PMID 27568074
- [Background] Filgueiras A, Hall CR. Psychometric properties of the Brazilian-adapted version of Sport Imagery Questionnaire. Psicol Reflex Crit. 2017 Oct 4;30(1):22. doi: 10.1186/s41155-017-0075-7. PMID 32025976